CLINICAL TRIAL: NCT01635101
Title: A Randomized, Placebo Controlled, Multi-Center Study of the Efficacy, Pharmacokinetics (PK) and Pharmacodynamics (PD) of IV Acetaminophen for the Treatment of Acute Pain in Pediatric Patients
Brief Title: A Multi-Center Study of the Efficacy, Pharmacokinetics (PK) and Pharmacodynamics (PD) of IV Acetaminophen for the Treatment of Acute Pain in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPI-APA-353
Record Dates: First submitted 2012-06-29; First posted 2012-07-06 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2017-05

CONDITIONS: Acute Pain
Keywords: Moderate to severe acute pain following surgery or trauma
MeSH Terms: conditions — Acute Pain; Wounds and Injuries | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Acetaminophen (Experimental): Participants receive a low dose of acetaminophen intravenously (IV) for 24 hours
  Interventions: Drug: IV Acetaminophen
- High Dose Acetaminophen (Experimental): Participants receive a low dose of acetaminophen (IV) for 24 hours
  Interventions: Drug: IV Acetaminophen
- Placebo (Placebo Comparator): Participants receive matching placebo (IV) for 24 hours
  Interventions: Drug: IV Control

INTERVENTIONS:
Drug: IV Acetaminophen — IV Acetaminophen given every 6 hours (q6h); 4 doses, in 24 hours
  Other Names: OFIRMEV
  Arms: High Dose Acetaminophen; Low Dose Acetaminophen
Drug: IV Control — IV Control q6h; 4 doses, in 24 hours
  Other Names: Saline; Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of Intravenous (IV) acetaminophen plus rescue opioids for the relief of moderate to severe acute pain in neonates and infants (age < 2 years) compared to placebo plus standard of care rescue opioids as well as characterize the concentration-effect relationship (PK/PD) of the intravenous acetaminophen as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 28 weeks gestational age and < 2 years old at study enrollment
* Subject will undergo surgery or had a traumatic injury expected to produce moderate to severe pain and patient is expected to require analgesic treatment for acute pain for 24 hours
* Subject has a medically reasonable need for IV treatment due to their underlying procedure(s) or medical condition(s) for the duration of the study
* Subject has reliable vascular access for administration of study medication and PK sampling
* Subject has a bodyweight which, in the opinion of the Investigator does not preclude participation in the study.
* Subject is free of other physical, mental, or medical conditions which, in the opinion of the Investigator, make study participation inadvisable or make it impossible to accurately assess efficacy or safety endpoints
* Subject's parent or guardian must provide written informed consent prior to participation in the study
* Subject's parent or guardian must have the ability to read and understand the study procedures and have the ability to communicate meaningfully with the study investigator and staff

Exclusion Criteria:

* Subject is not able to comply with the sampling requirements of the study
* Subject has known or suspected hypersensitivity to acetaminophen or the excipients of IV acetaminophen
* Subject has any significant medical condition that in the opinion of the Investigator contraindicates participation in the study or impairs the assessment of efficacy or safety
* Subject has participated in another interventional clinical study within 30 days of the planned study randomization date

Pre-Randomization (Qualification) Inclusion Criteria

Subject has not been administered any of the following:

* any acetaminophen-containing product, nonsteroidal anti-inflammatory agent, central alpha-adrenergic agents (e.g., clonidine, dexmedetomidine) or ketamine within 6 hours of baseline (T0)
* received a regional or neuraxial (caudal, epidural or spinal) anesthetic with local anesthetics within 6 hours of T0
* Subject does not have abnormal liver function tests from a sample obtained post-operatively/post-trauma and prior to randomization above protocol-specified limits
* Subject does not have significantly impaired renal function or known significant renal disease which in the opinion of the Investigator would contraindicate study participation.
* Subject had a nursing assessment documenting moderate to severe pain within 6 hours prior to randomization
* Subject required at least one dose of parenteral opioid medication for pain management (i.e., not pre-emptive therapy) during the 6-hour pre-randomization period, and is anticipated to require at least one dose of parenteral opioid medication during the 24 hour treatment period
* If subject is breast feeding, mother has not been administered any acetaminophen containing product in the previous 6 hours to T0 and throughout the treatment period

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (22):
- United States (22):
  - Children's Of Alabama, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hosptial San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Jackson Memorial Hospital, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Amplatz Children's Hospital, Minneapolis, Minnesota
  - Kings County Hospital Center, Brooklyn, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Univ. of Texas Health Sciences Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammer GB, Maxwell LG, Taicher BM, Visoiu M, Cooper DS, Szmuk P, Pheng LH, Gosselin NH, Lu J, Devarakonda K. Randomized Population Pharmacokinetic Analysis and Safety of Intravenous Acetaminophen for Acute Postoperative Pain in Neonates and Infants. J Clin Pharmacol. 2020 Jan;60(1):16-27. doi: 10.1002/jcph.1508. Epub 2019 Aug 25. PMID 31448420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 215 participants screened, 197 were actually enrolled and received study drug
Groups:
- Low Dose Acetaminophen: Participants receive a low dose of acetaminophen for 24 hours
- High Dose Acetaminophen: Participants receive a high dose of acetaminophen for 24 hours
- Placebo: Participants receive matching placebo administered intravenously for 24 hours
Period: Overall Study
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Started | 61 | 67 | 69
Safety Population | 61 | 67 | 69
Modified Intent to Treat (mITT) | 61 | 67 | 69
Pharmacokinetics Evaluable Population | 50 | 59 | 58
Completed | 52 | 55 | 52
Not Completed | 9 | 12 | 17

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population
Groups:
- Low Dose Acetaminophen: Participants received a low dose of acetaminophen for 24 hours
- Placebo: Participants receive matching placebo for 24 hours
- Total: Total of all reporting groups
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo | Total
Number analyzed (Participants) | 61 | 67 | 69 | 197
Age, Customized [Count of Participants; unit: Participants]
  All Participants: Neonates (birth to ≤ 28 days) | 13 | 12 | 13 | 38
  All Participants: Younger infants (≥ 29 days to < 6 mos) | 16 | 20 | 18 | 54
  All Participants: Intermediate aged infants (≥ 6 mos to <12 mos) | 18 | 17 | 20 | 55
  All Participants: Older infants (≥12 mos to <24 mos) | 14 | 18 | 18 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 27 | 26 | 70
  Male | 44 | 40 | 43 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 4 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 9 | 30
  White | 40 | 49 | 46 | 135
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 61 | 67 | 69 | 197

OUTCOME MEASURES:

1. Primary Outcome: Total Rescue Opioid Consumption
Description: Total micrograms per kilogram (µg/kg) of rescue opioid used during the same 24 hours the subject is on study medication
Time Frame: in 24 hours
Population: mITT population
Measure: Mean (Standard Deviation); unit: µg/kg
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 61 | 67 | 69
µg/kg | 166.9 (225.06) | 179.9 (193.47) | 180.2 (184.70)
Statistical Analysis 1: Comparison: Low Dose Acetaminophen vs Placebo; Difference in Least Squares (LS) Means; Test type: Other; p = 0.736, ANOVA; LS Mean Difference = -11.8, 97.5% CI 2-sided [-91.0 to 67.3]
Statistical Analysis 2: Comparison: High Dose Acetaminophen vs Placebo; LS Mean Difference; Test type: Other; p = 0.967, ANOVA; LS Mean Difference = 1.4, 97.5% CI 2-sided [-75.9 to 78.7]

2. Secondary Outcome: Time to First Rescue Medication
Time Frame: within 24 hours
Population: mITT population
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Low Dose Acetaminophen: Participants receive low dose acetaminophen for 24 hours
- High Dose Acetaminophen: Participants receive high dose acetaminophen for 24 hours
- Placebo: Participants receive placebo for 24 hours
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 61 | 67 | 69
hours | 4.78 [3.15 to 16.32] | 4.76 [2.15 to 10.08] | 3.81 [2.25 to 8.95]

3. Secondary Outcome: Summary of Pain Intensity Using the Leuven Neonatal Pain Scale (LNPS) in Neonates
Description: The LNPS is used for assessing pain intensity in neonates. Scores on the scale run from 0-14. Higher scores mean worse pain.
Time Frame: within 24 Hours
Population: Neonates in the mITT population with scores at each data collection time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 13 | 12 | 13
score on a scale
  at 0 hours | 0.8 (1.09) | 0.8 (1.27) | 1.1 (1.26)
  at 6 hours | 1.1 (1.04) | 1.0 (1.41) | 1.2 (1.82)
  at 12 hours | 2.2 (1.92) | 1.8 (1.76) | 2.0 (1.83)
  at 18 hours | 1.0 (1.53) | 1.8 (1.99) | 0.8 (0.99)
  at 24 hours: number analyzed (Participants) | 12 | 12 | 13
  at 24 hours | 0.8 (1.40) | 1.3 (1.42) | 0.9 (1.40)

4. Secondary Outcome: Summary of Pain Intensity Using the LNPS in Younger Infants
Description: The LNPS is used for assessing pain intensity in younger infants. Scores on the scale run from 0-14. Higher scores mean worse pain.
Time Frame: within 24 hours
Population: Younger Infants in the mITT population with scores at each data collection time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 16 | 20 | 18
score on a scale
  at 0 hours | 2.1 (2.85) | 1.5 (1.85) | 2.2 (2.05)
  at 6 hours: number analyzed (Participants) | 16 | 18 | 17
  at 6 hours | 2.1 (2.36) | 1.3 (1.33) | 2.4 (3.10)
  at 12 hours: number analyzed (Participants) | 16 | 18 | 16
  at 12 hours | 2.2 (2.4) | 1.8 (1.58) | 1.9 (1.24)
  at 18 hours: number analyzed (Participants) | 16 | 15 | 14
  at 18 hours | 1.6 (2.25) | 1.7 (2.06) | 2.1 (1.44)
  at 24 hours: number analyzed (Participants) | 14 | 15 | 14
  at 24 hours | 2.3 (1.59) | 1.3 (1.63) | 2.9 (2.51)

5. Secondary Outcome: Pain Intensity Using the FLACC Score in Intermediate Aged Infants
Description: The Face, Leg, Activity, Cry, and Consolability (FLACC) scale is used to assess pain intensity in intermediate aged infants. The scale is scored in a range of 0-10 with 0 representing no pain. A higher score means more pain.
Time Frame: within 24 hours
Population: Intermediate aged infants in the mITT population with a score at each data collection time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 18 | 17 | 20
score on a scale
  at 0 hours: number analyzed (Participants) | 15 | 17 | 18
  at 0 hours | 0.6 (1.30) | 1.6 (2.27) | 1.2 (2.05)
  at 6 hours: number analyzed (Participants) | 14 | 17 | 15
  at 6 hours | 0.7 (0.83) | 2.1 (2.71) | 1.4 (2.59)
  at 12 hours: number analyzed (Participants) | 13 | 17 | 12
  at 12 hours | 1.2 (1.41) | 0.08 (1.39) | 1.8 (2.49)
  at 18 hours: number analyzed (Participants) | 11 | 15 | 13
  at 18 hours | 1.4 (2.01) | 0.9 (1.19) | 0.5 (0.97)
  at 24 hours: number analyzed (Participants) | 11 | 14 | 12
  at 24 hours | 1.4 (2.29) | 0.9 (1.56) | 0.3 (0.65)

6. Secondary Outcome: Pain Intensity Using the FLACC Score in Older Infants
Description: The FLACC scale is used to assess pain intensity in older infants. The scale is scored in a range of 0-10 with 0 representing no pain. A higher score means more pain.
Time Frame: within 24 hours
Population: Older infants in the mITT population with a score at each data collection time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
Number analyzed (Participants) | 14 | 18 | 18
score on a scale
  at 0 hours: number analyzed (Participants) | 14 | 18 | 17
  at 0 hours | 2.2 (2.64) | 1.8 (2.65) | 1.8 (2.37)
  at 6 hours: number analyzed (Participants) | 12 | 16 | 15
  at 6 hours | 0.5 (0.90) | 1.2 (2.07) | 1.5 (2.42)
  at 12 hours: number analyzed (Participants) | 12 | 15 | 14
  at 12 hours | 0.8 (1.27) | 1.7 (2.76) | 2.4 (1.78)
  at 18 hours: number analyzed (Participants) | 10 | 14 | 14
  at 18 hours | 1.3 (1.95) | 0.1 (0.36) | 1.3 (2.67)
  at 24 hours: number analyzed (Participants) | 12 | 14 | 12
  at 24 hours | 2.0 (2.59) | 0.8 (1.12) | 0.1 (0.29)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Low Dose Acetaminophen | High Dose Acetaminophen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/67 | 2/69
Other Adverse Events (participants affected / at risk) | 21/61 | 8/67 | 24/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Acetaminophen (N=61) | High Dose Acetaminophen (N=67) | Placebo (N=69)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Leucocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Acetaminophen (N=61) | High Dose Acetaminophen (N=67) | Placebo (N=69)
Tachycardia (Cardiac disorders) | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 7 | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 2 | 2
Pyrexia (General disorders) | 3 | 3 | 13
Body temperature increased (Investigations) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure of individual investigator/site results is restricted for 18 months after final evaluation of study results or after release of a cooperative publication including all study from all sites, whichever occurs first. The sponsor has 60 days to review and comment on the publication and can request removal of any confidential information prior to public disclosure or publication.